CLINICAL TRIAL: NCT04868318
Title: The Impact of Intervention With High-protein Pre-digested Enteral Formula on Clinical Outcomes in Surgical Critically Ill Patients.
Brief Title: The Impact of Intervention With High-protein Enteral Formula in SICU.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tungs' Taichung Metroharbour Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 109067
Record Dates: First submitted 2021-04-22; First posted 2021-04-30 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Enteral Nutrition; Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VHP(very-high protein) group (Experimental): In VHP(very-high protein) group, we will provide pre-digested formula of 37% protein to the experimental group for at least 3 days to up to 7 days.
  Interventions: Other: Very-high protein enteral formula
- SHP(standard-high protein) group (Active Comparator): SHP(standard-high protein) group is the control group, standard-high protein formula (16% of energy) would be given to the control group for at least 3 days to up to 7 days.
  Interventions: Other: Standard-high protein enteral formula

INTERVENTIONS:
Other: Very-high protein enteral formula — Peptamen® Intense VHP (37% protein)
  Arms: VHP(very-high protein) group
Other: Standard-high protein enteral formula — Peptamen® (16% protein)
  Arms: SHP(standard-high protein) group

SUMMARY:
The advantage of higher protein intake has been pointed for critically ill patients. However, it is not easy to achieve no overfeeding but adequate protein intakes for critically ill patients. It is thus important to conduct a strategy to deliver an adequate protein under but no overfeeding for critically ill patients. The purpose of this study is to investigate the association of protein intakes with clinical outcomes by delivering high-protein pre-digested enteral formula to surgical critically ill patients. We are going to recruit 160 surgical critically ill patients. Patients would be randomly assigned to either control or experimental group. Very-high protein pre-digested formula (37% of energy) would be given to the experimental group, while standard-high protein formula (16% of energy) would be given to the control group for at least 3 days to up to 7 days. The patients' data were collected or calculated and included basic characteristics, mean energy and protein intakes, clinical outcomes (APACHE II score, comorbidities, days in hospital to ICU admission, length of ventilator dependence, hospital and ICU stays, and survival days). We anticipated that the results of this study could provide the benefit of high protein delivery on clinical outcomes for critically ill patients.

DETAILED DESCRIPTION:
Trial Design and Patient Population

This study is an investigator-initiated, prospective, randomized controlled trial. This study is conducted according to the guidelines laid down in the Declaration of Helsinki, and all procedures were reviewed as well as approved by the Regional Hospital Ethics Committee. The written informed consent will be obtained before randomization. We will collect subjects' demographic and clinical characteristics on the first and seventh day of the intervention, including age, gender, weight, height, body mass index (BMI), Disease diagnosis, disease severity (The Acute physiology and Chronic Health Evaluation II, APACHE II), Sequential Organ Failure Assessment (SOFA) Score, disease history, ventilator parameters, body temperature, blood pressure, pulse rate and breathing frequency. The complications, length of stay in intensive care unit, total hospitalization Days, hospital mortality, 14-day survival results, 28-day survival results, days of ventilator use will be also recorded.

Patients 20 years of age or older will be eligible for inclusion if they have been admitted to the surgical Intensive Care Unit (SICU) for 24 hours or more. Subjects with enteral nutrition to be clinically contraindicated by treating clinician considered will be excluded. Total of one hundred and sixty patients will be included and randomly assigned into two groups.

Anthropometric and Biochemical Assessments

The patients' caloric requirement will be calculated based on the guidelines for critically ill nutrition treatment published by ASPEN/SCCM in 2016, suggesting that critically ill patients should be given 25 calories per kilogram of ideal body weight. The protein requirement of patients will be calculated based on the 1.5 g/kg/day recommended by the 2017 ESPEN guidelines for the nutritional care of critically ill surgical patients.

The nutritional intake and digestive tract symptoms of the patient within 7 days after entering the intensive care unit will be recorded, including nutritional intake (calories, carbohydrate, protein, fat) of enteral nutrition as well as intravenous nutrition(dosage of propofol, glucose infusion and glucosaline used...etc.),and digestive symptoms (diarrhea, bloating, Abdominal pain, constipation, nausea, vomiting... etc.).

The biochemical assessments of patients will be measured on the first and seventh days of admission to the ICU, including blood routine examination, total lymphocyte counts, creatinine, blood urine nitrogen, alanine aminotransferase (ALT), aspirate aminotransferase (AST), total bilirubin, albumin, prealbumin, total protein, cholesterol, triglyceride, uric acid, electrolyte, C-reactive protein, blood sugar as well as 24-hour urine urea nitrogen (UUN).

Total Lymphocyte Count and Nitrogen Balance are calculated by the following formulae.

Total Lymphocyte Count (cells/mm3) = WBC×% lymphocyte Nitrogen Balance (gm/day) = (protein intake/6.25) - (UUN + 4 g obligatory loss)

Intervention Formula In-kind support will be provided by Nestlé Health Science, which supplied both of the enteral nutrition formulations, Peptamen® Intense VHP and Peptamen®. Peptamen® Intense VHP (37% protein of total energy) and Peptamen® (16% protein of total energy) will be provided to two groups of subjects respectively.

The trial enteral nutrition was administered for at least 3 days up to 7 days or until the patient discontinued enteral nutrition, or was discharged from the ICU, whichever occurred first.

ELIGIBILITY:
Inclusion Criteria:

* 20 years of age or older.
* Those who have stayed in the surgical intensive care unit for 24 hours or more.

Exclusion Criteria:

* Those who cannot supply enteral nutrition within 3 days due to disease or unstable clinical conditions.
* Those who have been fed for less than three days due to disease or unstable clinical conditions.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Survival rate | 28 days
  The percentage of people in two-arm group was still alive for 28-days of time after admission to ICU.
Survival rate | 14 days.
  The percentage of people in two-arm group was still alive for 14-days of time after admission to ICU.

SECONDARY OUTCOMES:
ICU days | 28 days
  ICU days is the duration of a single episode of ICU. It is calculated by subtracting day of ICU admission from day of ICU discharge.
Hospital days | 28 days
  Hospital days, be equal length of stay (LOS), is the duration of a single episode of hospitalization. It is calculated by subtracting day of admission from day of discharge.
Length of ventilator | 28 days
  Length of ventilator is the total days of using ventilator. It is calculated by recording whether ventilator was used on the day in ICU.
Nitrogen balance | 7 days
  Nitrogen balance, calculated by measuring urine urea nitrogen (UUN) to assess whether the protein state is sufficient.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Rong Li, Principal Investigator — Tungs' Taichung Metroharbor Hospital; Yi-Chia Huang, Principal Investigator — Chung Shan Medical University; Shung-Sheng Tsou, Principal Investigator — Tungs' Taichung Metroharbor Hospital; Li-Wa Liao, Study Director — Tungs' Taichung Metroharbor Hospital; Feng-Chan Shi, Study Chair — Tungs' Taichung Metroharbor Hospital
Locations (1):
- PS Lim, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No